CLINICAL TRIAL: NCT00549393
Title: Impact of Daily Bathing With Chlorhexidine Impregnated Cloths on Nosocomial Infections in the Pediatric Intensive Care Unit
Brief Title: Study of Bathing With Chlorhexidine Impregnated Cloths on Nosocomial Infections in the Pediatric Intensive Care Unit
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Sage Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NA_00006799
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Nosocomial Infections
Keywords: intensive care unit; Healthcare associated infections (HAI); pediatric
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Daily bathing with 2% chlorhexidine gluconate
  Interventions: Drug: 2% Chlorhexidine gluconate cloth
- 2 (No Intervention): Standard bathing with soap and water basin or disposable cloth

INTERVENTIONS:
Drug: 2% Chlorhexidine gluconate cloth — Daily bathing
  Arms: 1

SUMMARY:
The investigators propose to conduct a large clinical study to determine if daily bathing with chlorhexidine impregnated cloths will reduce the incidence of healthcare-associated infections in the Pediatric Intensive Care Unit (PICU).

ELIGIBILITY:
Inclusion Criteria:

* Patients in pediatric intensive care unit

Exclusion Criteria:

* Patients with a history of an allergic reaction to chlorhexidine
* Patients less than 2 months of age
* Patients with severe skin disease or burn
* Patients with an indwelling epidural catheter or lumbar drain

Ages: 2 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5659 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trish M Perl, MD MSc, Principal Investigator — Johns Hopkins University; Aaron Milstone, MD MHS, Study Chair — Johns Hopkins University
Locations (5):
- United States (5):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Result] Milstone AM, Elward A, Song X, Zerr DM, Orscheln R, Speck K, Obeng D, Reich NG, Coffin SE, Perl TM; Pediatric SCRUB Trial Study Group. Daily chlorhexidine bathing to reduce bacteraemia in critically ill children: a multicentre, cluster-randomised, crossover trial. Lancet. 2013 Mar 30;381(9872):1099-106. doi: 10.1016/S0140-6736(12)61687-0. Epub 2013 Jan 28. PMID 23363666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The hospital ICU units underwent a crossover study design, so the ICUs recruited participants in the assigned treatment or control group, then the unit had a washout period, then the unit switched to the alternative assignment of intervention or control for a separate population of participants that were admitted into the ICU.
Pre-assignment Details: 5659 enrolled visits in the study, but 712 were excluded from analysis as they did not meet the eligibility criteria
Groups:
- 2% Chlorhexidine Gluconate Cloth: Daily bathing with 2% chlorhexidine gluconate
  2% Chlorhexidine gluconate cloth: Daily bathing
- Standard Bath: Standard bathing with soap and water basin or disposable cloth
Period: Period 1 (6 Months)
Arm/Group | 2% Chlorhexidine Gluconate Cloth | Standard Bath
Started | 1319 (intention to treat (ITT)) | 1199 (ITT)
Per Protocol | 880 | 1199
Completed | 1319 | 1199
Not Completed | 0 | 0
Period: Period 2 Washout (2 Weeks)
Arm/Group | 2% Chlorhexidine Gluconate Cloth | Standard Bath
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0
Period: Period 3 (6 Months)
Arm/Group | 2% Chlorhexidine Gluconate Cloth | Standard Bath
Started | 1103 (number not equal to period 1 due to unit cross over design) | 1326 (number not equal to period 1 due to unit cross over design)
Per Protocol | 667 | 1326
Completed | 1103 | 1326
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Daily bathing with 2% chlorhexidine gluconate
  2% Chlorhexidine gluconate cloth: Daily bathing
- Control Arm: Standard bathing with soap and water basin or disposable cloth
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 2422 | 2525 | 4947
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 4.8 [1.1 to 12.9] | 4.8 [1.1 to 12.7] | 4.8 [1.1 to 12.9]
Sex/Gender, Customized [Number; unit: participants]
  Male | 1389 | 1388 | 2777
  Female | 1033 | 1137 | 2170
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1271 | 1269 | 2540
  non-Caucasian | 1151 | 1256 | 2407
PRISM III Score [Median (Inter-Quartile Range); unit: score] — Severity score that predicts mortality. Range 0 (lowest mortality risk) to 74 (highest mortality risk)
  score | 5 [0 to 13] | 5 [0 to 11] | 5 [0 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Bacteremia
Description: incidence of bacteremia comparing those in treatment and control groups
Time Frame: participants were followed for the duration of ICU stay, median stay 3 days
Population: Intent to treat population
Measure: Number (95% Confidence Interval); unit: events per 1000 at-risk days
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 2422 | 2525
events per 1000 at-risk days | 3.52 [2.64 to 4.61] | 4.93 [3.91 to 6.15]

2. Secondary Outcome: Central Line Associated-bloodstream Infection (CLABSI)
Description: Comparing incidence of central line-associated bloodstream infections between treatment and control groups
Time Frame: participants were followed for the duration of ICU stay, median stay 3 days
Measure: Number (95% Confidence Interval); unit: events per 1000 at-risk days
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 2422 | 2525
events per 1000 at-risk days | 1.63 [0.87 to 2.79] | 3.00 [2.00 to 4.33]

3. Other Pre Specified Outcome: Bacteremia
Description: per protocol analysis of incidence of bacteremia comparing those in treatment and control groups
Time Frame: duration of ICU stay, median 3 days
Population: Includes per protocol population of 1547 of 2422 in the treatment arm
Measure: Number (95% Confidence Interval); unit: events per 1000 at-risk days
Groups:
- Treatment: Daily bathing with 2% chlorhexidine gluconate
- Control: Standard bathing with soap and water basin or disposable cloth
Arm/Group | Treatment | Control
Number analyzed (Participants) | 1547 | 2525
events per 1000 at-risk days | 3.28 [2.277 to 4.58] | 4.93 [3.91 to 6.15]

ADVERSE EVENTS:
Time Frame: participants were followed for the duration of ICU stay, median stay 3 days
Arm/Group | Treatment Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/2422 | 0/2525
Other Adverse Events (participants affected / at risk) | 43/2422 | 26/2525
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=2422) | Control Arm (N=2525)
Skin reaction (Skin and subcutaneous tissue disorders) | 43 (43) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No